CLINICAL TRIAL: NCT00350428
Title: Angle Closure: Laser Iridotomy Versus Phacoemulsification Study (ACLIPS)- A Study of Acute Primary Angle Closure Glaucoma Comparing Two Treatment Modalities: Laser Peripheral vs Phacoemulsification With Posterior Intraocular Lens Implant
Brief Title: Laser Iridotomy Versus Phacoemulsification in Acute Angle Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R221/13/2001; SQGL05
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2004-10

CONDITIONS: Angle Closure Glaucoma
Keywords: Acute primary angle closure; Laser preipheral iridotomy; Phacoemulsification
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Phacoemulsification

INTERVENTIONS:
Procedure: Laser Preipheral Iridotomy and phacoemulsification

SUMMARY:
This is a randomised controlled clinical trial to compare laser peripheral iridotomy (LPI) and primary phacoemulsification with intra-ocular lens implantation (phaco/IOL) in the treatment of acute primary angle-closure glaucoma (APACG). Following successful medical lowering of raised intra-ocular pressure (IOP) and control of intraocular inflammation, patients presenting to Singapore National Eye Centre and Singapore General Hospital with acute primary angle-closure glaucoma who meet the eligibility are randomised to one of the two treatment arms: laser peripheral iridotomy and primary phacoemulsification with intra-ocular lens implantation. These patients will be monitored closely for 2 years post-operatively.

DETAILED DESCRIPTION:
AIMS

The objective of this study is to conduct a randomised controlled clinical trial to compare LPI and primary phacol/IOL in the treatment of APACG.

The specific aim is to compare long-term IOP control in patients who undergo LPI with patients who undergo primary phaco/IOL. At the same time the following will be studied.

1. To evaluate the safety of these two techniques for the treatment of APACG
2. To assess the development of PAS
3. To establish if LPI and primary phaco/IOL are as effective in preventing the recurrence of acute attack in eyes with APACG

TREATMENT PLAN

Initial Medical Treatment

Patients with APACG will be treated initially for the acute attack with medical treatment. The initial treatment is standardized to the following:

1. Intravenous acetazolamide (Diamox) 500 mg stat
2. Oral acetazolamide 250 mg tid to qid with Span K 1.2 g om
3. Topical beta-blocker (Timolol 0.5%) bid or Brimonidine bid if beta-blockers are contra-indicated.
4. Topical pilocarpine 4% qid
5. Topical steroids
6. Intravenous mannitol 20% at 1-2g/kg at 4 hours after initiation of treatment if IOP is not reduced by 20% of initial IOP unless contra-indicated due to systemic disease eg. Congestive heart failure.
7. A second infusion of intravenous mannitol 20% at 2g/kg at 12 hours after initiation of treatment if IOP is still not reduced by 20% of initial IOP

Response to Initial Treatment and Evaluation of Cataract

Patients are divided into 2 categories based on IOP after 24 hours of initiation of medical treatment: (a) APACG with IOP £ 30 mmHg (b) APACG with IOP > 30 mmHg.

Patients with IOP £ 30 mmHg are evaluated clinically for the presence of cataract and further divided into those with cataract and those without cataract. Patients with cataract are defined as those with best corrected visual acuity equal or less than 6/15 due to lens opacity in the opinion of a consultant grade ophthalmologist.

Note: Eyes with intumescent cataract (phacomorphic glaucoma), subluxated lens or anterior chamber depth differing by more than 0.3 mm are excluded.

Eligible patients with informed consent are randomised.

Laser Peripheral Iridotomy

1. In addition to the consultants, LPI may be performed by registrars, senior registrars and fellows who have observed and been taught by the glaucoma consultants and are deemed to be able to perform the procedure to a high standard.
2. LPI is performed when the cornea is sufficiently clear (usually within 72 hours) following the lowering of the IOP medically.
3. Technique for LPI to be standardized to sequential argon-Nd-YAG Laser PI.
4. LPI should be sited at the superior nasal or superior temporal quadrant.
5. The size of opening should be ³ 200mm.
6. Following successful LPI, topical eyedrops are continued for one week after the procedure. Oral Diamox is discontinued.
7. If the initial attempt is unsuccessful, LPI at a second alternative site will be attempted. If the second attempt remains unsuccessful, patient will be considered as failure .

Phacoemulsification with Intra-ocular Lens Implantation

1. All phacoemulsification with intraocular lens implantation are to be performed by consultant surgeons. The panel of surgeons is formed from the group of co-investigators of this study.
2. Phacoemulsification will be carried out between 5 to 7 days following the lowering of the IOP. This is to allow for improved corneal clarity and reduction of intra-ocular inflammation.
3. Gutt pilocarpine to be stopped on morning of operation.
4. Pre-operative intravenous mannitol 20% at 1-2g/kg is given 2 hours before the start of operation for those subjects with an IOP persistently raised above 21mmHg.
5. Clear corneal incision.
6. Viscoelastic agent to be injected 360 degrees circumferentially in the angles to deepen the anterior chamber. There will be no other angle augmentation procedure using surgical instruments.
7. A standard foldable IOL (Type of IOL: Acrysof MA60)
8. Viscoelastic agent should be removed at the end of operation as far as possible.
9. Oral Diamox 250 mg to be given stat post-operatively to reduce post-operative IOP spike.
10. Following successful phacoemulsification with IOL implantation, topical steroids and antibiotics are given. Topical pilocarpine, timolol and oral Diamox are stopped.

IOP Lowering Medication

With regard to the determination of endpoints IOP evaluation will be considered from post-operative week 3 onward. This is to allow for treatment of short-term surgery related IOP fluctuation.

During the follow up period, if a rise of IOP occurs, i.e. IOP is between 22 to 24 mmHg on two occasions within one month or IOP ³ 25 mmHg on one occasion, IOP lowering medication will be started.

FOLLOW-UP

Post operation visit Window period

1st week ± 2 days 3rd week ± 5 days 6th week ± 7 days 3rd month ± 2 weeks 6th month to 2nd year ± 3 weeks

At the completion of the trial patient will receive normal clinical follow up of 4-6 monthly thereafter whilst the data will not be collected for this study.

The primary objective of the study is to compare IOP control between these two treatment groups.

STATISTICAL CONSIDERATIONS

Sample Size Calculation:

The primary objective of the study is to compare long-term intra-ocular pressure (IOP) control between the two groups.

The proportion of the subjects whose IOP are not successfully controlled in the LPI group can be estimated as 60% (Aung T 2001). And the proportion of the subjects whose IOP are not successfully controlled in the phacoemulsification with intra-ocular lens implant group is about 20% under clinical estimation. Hence, the study needs a sample size of 70 patients (Machin, Campbell, Fayers & Pinol, 1997), 35 in each group. This will be sufficient to detect a 60% vs. 20% of proportion of the subjects who develop increasing IOP between two groups with a two-sided test with a power 90% while the significance level is controlled at 5%.

Statistical Analysis Plan

All statistical analysis will be carried out on an intention-to-treat basis. In the event of lost to follow-up, patients will still be included in the analysis for the duration that they are observed, and the last IOP which is assessed before lost to follow-up will be used for data analysis.

To compare long-term IOP control between two treatments, Pearson χ2 test or Fisher's exact test will be used. The evaluation of the incidence of recurrence of an acute attack in eyes with APACG will be carried out using Fisher's exact test. Logistic regression will be carried out to adjust for relevant covariates.

The time interval for the subsequent increase in IOP to occur after LPI or phacol/IOL is to be recorded. Kaplan-Meier life table analysis can be applied to assess the survival time (failure being defined as any need for further glaucoma treatment) of two groups, and Log rank test will be used to compare the two survival curves. In addition, The Cox regression will be used to adjust for covariates where applicable.

An interim statistical analysis will be carried out after all patients have completed 6 months follow-up.

REFERENCES

1. Acton J, Salmon JF, Scholtz R. Extracapsular cataract extraction with posterior chamber lens implantation in primary angle-closure glaucoma. J Cataract Refract Surg. 1997 Jul-Aug;23(6):930-4.
2. Aung T, Ang LP, Chan SP, Chew PT. Acute primary angle-closure: long-term intraocular pressure outcome in Asian eyes. Am J Ophthalmol. 2001;131(1):7-12.
3. Chylack LTJ, Wolfe JK, Singer DM, et al. The Lens Opacities Classification System III. Arch Ophthalmol 1993;111:831-836.
4. Fleiss JL. Statistical methods for rates and proportions. New York:Wiley, 1981:2nd edition.
5. Greve EL Primary angle closure glaucoma: extracapsular cataract extraction or filtering procedure? Int Ophthalmol. 1988;12(3):157-62.
6. Gunning FP, Greve EL. Uncontrolled primary angle closure glaucoma: results of early intercapsular cataract extraction and posterior chamber lens implantation. Int Ophthalmol. 1991 Jul;15(4):237-47.
7. Gunning FP, Greve EL. Lens extraction for uncontrolled angle-closure glaucoma: long-term follow-up. J Cataract Refract Surg. 1998 Oct;24(10):1347-56.
8. Ho T, Fan R. Sequential argon-Yag laser iridotomies in dark irides. Br J Ophthalmol 1992; 76:329 -331.
9. Hoffer KJ. Axial dimensions of the human cataractous lens. Arch Ophthalmol 1993; 111(7):914-8.
10. Hong C, Kitazawa Y, Tanishima H. Influence of argon laser treatment of glaucoma on corneal endothelium. Japan J Ophthalmol 1983;27(4):567-74.
11. Ishikawa H, Ritch R, Liebmann J. Quantitative assessment of the anterior segment using Ultrasound Biomicroscopy. Current Opinions In Ophthalmology. 2000;11:133-139.
12. Lim L, Seah SKL, Lim ASM. Comparison of argon laser iridotomy and sequential argon laser and Nd:YAG laser iridotomy in dark irides. Ophthalmic surgery and lasers 1996;27(4):92-95.
13. Lowe RF. Aetiology of the anatomical basis for primary angle-closure glaucoma:biometrical comparisons between normal eyes and eyes with primary angle-closure glaucoma. Br J Ophthalmol 1970; 54(3):161-9.
14. Lowe RF: Primary angle-closure glaucoma: a review of ocular biometry, Aust NZ J Ophthalmol 1977; 5:9.
15. Lowe RF. Clinical types of primary angle-closure glaucoma. Aust NZ J Ophthalmol 1988;16:245-50.
16. Obstbaum SA. Glaucoma and intraocular lens implantation. J Cataract Refract Surg 1986;12:257-61.
17. Pavlin,CJ, Foster,FS. Ultrasound biomicroscopy in glaucoma. [Review]. Acta Ophthalmologica - Supplement. 1992;7-9.
18. Roberts TV, Francis IC, Lertusumitkul S, Kappagoda MB, Coroneo MT. Primary phacoemulsification for uncontrolled angle-closure glaucoma. J Cataract Refract Surg 2000;26:1012-16.
19. Teekhasaenee C, Ritch R. Combined phacoemulsification and goniosynechialysis for uncontrolled chronic angle-closure glaucoma after acute angle-closure glaucoma. Ophthalmology. 1999 Apr;106(4):669-74.
20. Wishart PK, Atkinson PL. Extracapsular cataract extraction and posterior chamber lens implantation in patients with primary chronic angle-closure glaucoma: effect on intraocular pressure control. Eye. 1989;3 ( Pt 6):706-12.

ELIGIBILITY:
Inclusion Criteria:

1. APACG. In cases where both eyes are eligible, the right eye will be entered.
2. IOP less than or equal to 30 mmHg within 24 hours of presentation and after initiation of medical treatment
3. Significant cataract with best corrected visual acuity equal or less than 6/15
4. Informed consent

Exclusion Criteria:

1. Secondary causes of angle-closure e.g. subluxed lens, uveitis, trauma and neovascular glaucoma
2. Intumescent cataract (phacomorphic glaucoma)
3. Eyes with anterior chamber depth differing by more than 0.3 mm
4. Eyes with no cataract
5. Active ocular infection in either eye which would prevent surgery
6. Female subjects who are pregnant, nursing or of childbearing potential and not using adequate contraception
7. Participating in another study
8. Previous intraocular eye surgery on the affected eye.
9. Any medical condition which would be a contra-indication to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2001-10; Study Completion 2007-10

PRIMARY OUTCOMES:
Recurrence of APACG: Patients who develop a recurrence of symptoms of APACG. Treatment of recurrence will be decided by the ophthalmologist managing the patient.
IOP lowering medication is required.
Further glaucoma surgery is required.

SECONDARY OUTCOMES:
Cataract surgery is required. Patients in the LPI group who develop significant progression of cataract during the follow-up period will be offered cataract extraction.
No light perception
Eyes become phthisical

CONTACTS AND LOCATIONS:
Overall Officials: Steve Seah, FRCS (Ed), Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore